CLINICAL TRIAL: NCT04693598
Title: A Phase 1/2 Clinical Study of Intravenous Gene Transfer With an AAVrh10 Vector Expressing GALC in Krabbe Subjects Receiving Hematopoietic Stem Cell Transplantation (RESKUE)
Brief Title: Gene Transfer Clinical Trial for Krabbe Disease
Acronym: RESKUE
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Forge Biologics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FBX-101-RESKUE
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Krabbe Disease
Keywords: Lysosomal Storage Disorder; Globoid Cell Leukodystrophy; Leukodystrophy; GALC
MeSH Terms: conditions — Leukodystrophy, Globoid Cell; Lysosomal Storage Diseases

STUDY DESIGN:
Intervention Model Description: Dose escalation study from a low dose to a high dose following safety review
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Low Dose FBX-101 (aka AAVrh.10-GALC) (Experimental): Participants will receive a single infusion at the lower dose (N=3 participants)
  Interventions: Biological: FBX-101
- Cohort 2 - High Dose FBX-101 (aka AAVrh.10-GALC) (Experimental): Participants will receive a single infusion at the higher dose (N=3 participants)
  Interventions: Biological: FBX-101

INTERVENTIONS:
Biological: FBX-101 — A replication-deficient adeno-associated virus gene transfer vector expressing the human galactocerebrosidase (GALC) cDNA will be delivered one-time through a venous catheter inserted into a peripheral limb vein.
  Other Names: AAVrh.10-hGALC

SUMMARY:
This is a nonblinded, non-randomized dose escalation study of intravenous AAVrh10 after hematopoietic stem cell transplantation (HSCT) in which subjects will receive standard of care hematopoietic cell transplantation for Krabbe disease, followed by a single infusion of an adeno-associated virus gene therapy product. Extensive natural history subjects will be used to compare as control group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of infantile Krabbe disease, characterized by the following criteria outlined below:

   * Galactocerebrosidase (GALC) activity levels in leukocytes compatible with the diagnosis of Krabbe disease; AND AT LEAST ONE OF THE FOLLOWING:
   * Elevated psychosine levels predictive of infantile disease onset by DBS; OR
   * Imaging or neurophysiological findings consistent with Krabbe disease (CSF, MRI, NCV, ABR); OR
   * Two GALC mutations predictive to result in infantile onset phenotype.
2. Age at the time of screening: 1 day to 12 months
3. Participant has been deemed eligible for treatment with HSCT (standard of care) and a fully myeloablative reduced intensity/toxicity conditioning regimen (RIC/RTC) is/has been used
4. Participant's parents or legal guardian consents to participate in the study and provides informed consent according to IRB guidelines prior to any study procedures being performed
5. Parent(s) and/or legal guardian able to comply with the clinical protocol
6. Participant must have adequate organ function at time of screening as measured by:

   * Creatinine ≤ 1.5x upper limit of age appropriate normal and creatinine clearance ≥ 60 mL/min/1.73 m2
   * Hepatic transaminases (ALT/AST) ≤ 2x age related upper limit of normal
   * Ejection fraction of > 50% by echocardiogram or other appropriate study without evidence of pulmonary hypertension
   * Pulmonary evaluation testing demonstrating resting pulse oximeter > 95% on room air
   * Coagulation tests within 110% of normal ranges for age. (PT/INR and PTT)

Exclusion Criteria:

1. History of prior treatment with a gene therapy product
2. Presence of major congenital anomaly or any other condition that affects neurodevelopmental function
3. Presence of any neurocognitive deficit or brain damage not attributable to Krabbe disease
4. Active aspiration
5. Signs of active infection or disease from cytomegalovirus, adenovirus or other viruses
6. HIV positive
7. Uncontrolled and progressive bacterial or fungal infection
8. Presence of any contraindication for MRI
9. Use of any investigational product prior to study enrollment or current enrollment in another study that involves clinical interventions
10. Any other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the PI, would preclude participation in the study
11. Ongoing veno-occlusive disease (VOD) as determined by liver ultrasound (moderate ascites and static or retrograde portal vein flow) the day before FBX-101 infusion.

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by incidence and severity of adverse events and serious adverse events that are attributed to FBX-101. | 24 months
Safety as assessed by HSCT incident of engraftment. | 24 months

SECONDARY OUTCOMES:
Efficacy as assessed by improvement of probability to achieve independent sitting compared to untreated patients or those receiving HSCT only. | 12 months and 24 months
Efficacy as assessed by improvement of gross motor function as measured by Peabody Developmental Motor Scale 2nd Edition (PDMS-2) above a functional age equivalent of 12 months compared to untreated patients or those receiving HSCT only | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Hospitals - Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data

REFERENCES:
- [Derived] Bradbury AM, Bagel J, Swain G, Miyadera K, Pesayco JP, Assenmacher CA, Brisson B, Hendricks I, Wang XH, Herbst Z, Pyne N, Odonnell P, Shelton GD, Gelb M, Hackett N, Szabolcs P, Vite CH, Escolar M. Combination HSCT and intravenous AAV-mediated gene therapy in a canine model proves pivotal for translation of Krabbe disease therapy. Mol Ther. 2024 Jan 3;32(1):44-58. doi: 10.1016/j.ymthe.2023.11.014. Epub 2023 Nov 11. PMID 37952085
- [Derived] Heller G, Bradbury AM, Sands MS, Bongarzone ER. Preclinical studies in Krabbe disease: A model for the investigation of novel combination therapies for lysosomal storage diseases. Mol Ther. 2023 Jan 4;31(1):7-23. doi: 10.1016/j.ymthe.2022.09.017. Epub 2022 Oct 4. PMID 36196048
- See also: Bascou, N., DeRenzo, A., Poe, M. & Escolar, M., 2018. A prospective natural history study of Krabbe disease in a patient cohort with onset between 6 months and 3 years of life. Orphanet Journal of Rare Diseases, pp. 1-17. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6083585/
- See also: Beltran-Quintero, M. et al., 2019. Early progression of Krabbe disease in patients with symptom onset between 0 and 5 months. Orphanet Journal of Rare Diseases, pp. 1-13. — https://pubmed.ncbi.nlm.nih.gov/30777126/
- See also: Bradbury, A. et al., 2018. AAVrh10 Gene Therapy Ameliorates Central and Peripheral Nervous System Disease in Canine Globoid Cell Leukodystrophy (Krabbe Disease). Human Gene Therapy, pp. 785-801. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6066194/
- See also: Escolar, M. et al., 2005. Transplantation of Umbilical-Cord Blood in Babies with Infantile Krabbe's Disease. The New England Journal of Medicine, pp. 2069-2081. — https://pubmed.ncbi.nlm.nih.gov/15901860/
- See also: Escolar, M. et al., 2016. Clinical management of Krabbe disease. Journal of Neuroscience Research, pp. 1118-1125. — https://pubmed.ncbi.nlm.nih.gov/27638597/
- See also: Rafi, M., Luzi, P. & Wenger, D., 2020. Conditions for combining gene therapy with bone marrow transplantation in murine Krabbe disease. BioImpacts, pp. 105-115. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7186542/
- See also: Bradbury et al. 2023.Combination HSCT and intravenous AAV-mediated gene therapy in a canine model proves pivotal for translation of Krabbe disease therapy. Molecular Therapy, November 2023:S1525-0016(23)00615-9. — https://pubmed.ncbi.nlm.nih.gov/37952085/